CLINICAL TRIAL: NCT04026685
Title: Maternal Haemodynamic Changes After Crystalloid Co-loading and Phenylephrine Versus Phenylephrine Alone During Spinal Anaesthesia for Elective Caesarean Delivery: a Double-blind, Randomised Controlled Trial Using the Non Invasive Cardiac Output Monitor StarlingTM SV.
Brief Title: Maternal Haemodynamic Changes After Crystalloid Co-loading and Phenylephrine Versus Phenylephrine Alone During Spinal Anaesthesia for Elective Caesarean Delivery
Acronym: NICOM-USB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-00866; qu18Buddeberg
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Maternal Haemodynamic Stability
Keywords: caesarean delivery; phenylephrine; spinal anaesthesia; vasopressor administration; pregnancy; non invasive cardiac output (CO) monitoring (NICOM)

STUDY DESIGN:
Intervention Model Description: double-blind, randomised controlled non-inferiority trial
Who Masked: Participant, Investigator
Masking Description: Investigator and participant cannot see to which study group the participant belongs. The person performing randomisation and fluid application will not be involved in the data collection and Analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine infusion only (Active Comparator): Phenylephrine infusion only
  Interventions: Drug: Phenylephrine infusion
- Phenylephrine infusion and Ringer-Acetate bolus (Active Comparator): Phenylephrine infusion and Ringer-Acetate bolus
  Interventions: Drug: Phenylephrine infusion and Ringer-Acetate bolus

INTERVENTIONS:
Drug: Phenylephrine infusion — continuous phenylephrine infusion started at a rate of 25mcg/min and titrated according to blood pressure
  Arms: Phenylephrine infusion only
Drug: Phenylephrine infusion and Ringer-Acetate bolus — continuous phenylephrine infusion started at a rate of 25mcg/min and titrated according to blood pressure plus crystalloid Ringer-Acetate co-loading bolus of 1000 mL
  Arms: Phenylephrine infusion and Ringer-Acetate bolus

SUMMARY:
Spinal anaesthesia is the anaesthetic technique of choice for elective caesarean delivery. Hypotension, a result of the decrease in systemic vascular resistance caused by spinal anaesthesia, is a frequent complication occurring in up to 80%. This study is to investigate fluid loading plus vasopressors to vasopressors alone to maintain stable maternal haemodynamics in elective caesarean delivery. The effect of the two methods (continuous prophylactic phenylephrine infusion with and without crystalloid co-loading) on maternal haemodynamics will be compared using the Starling SV Monitor. The Starling SV device is a non invasive cardiac output monitor (NICOM) which is certified and validated for the use in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Term uncomplicated singleton pregnancy
* Undergoing elective caesarean section under spinal anaesthesia
* Weight: 50-100kg
* Height: 150-180cm
* Healthy term fetus

Exclusion Criteria:

* Inability to give informed consent
* Multiple pregnancy
* Clinically significant concomitant disease states (e.g. hypertension, cardiac disease, severe asthma requiring regular medication, comorbidities affecting the autonomous nervous system, renal disease)
* On any cardiovascular medication
* Complications of pregnancy (e.g. preeclampsia, intrauterine growth restriction, fetal malformations)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Any fetal pathology (e.g. fetal malformations, rupture of membranes before caesarean section, oligohydramnios, polyhydramnios, suspected chorioamnionitis)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2021-02-05 (Actual)

PRIMARY OUTCOMES:
Change in maternal cardiac output (CO) | measured every minute after induction of spinal anaesthesia (=baseline) until 5 minutes after cord clamping
  CO measured by area under the curve (AUC) (L/min.)

SECONDARY OUTCOMES:
Change in maternal heart rate | measured every minute after induction of spinal anaesthesia (=baseline) until 5 minutes after cord clamping
  Change in maternal heart rate
Change in maternal diastolic and systolic blood pressure | measured every minute after induction of spinal anaesthesia (=baseline) until 5 minutes after cord clamping
  Change in maternal diastolic and systolic blood pressure (mmHg)
incidence of maternal nausea | measured every minute after induction of spinal anaesthesia (=baseline) until 5 minutes after cord clamping
  incidence of maternal Nausea (number)
Change in Apgar scores | at 1 and 5 minutes after delivery
  The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form a backronym (Appearance, Pulse, Grimace, Activity, Respiration).
Change in umbilical cord pH | at 1 and 5 minutes after delivery
  Change in umbilical cord pH

CONTACTS AND LOCATIONS:
Overall Officials: Bigna Buddeberg, Dr. med, Principal Investigator — Department of Anaesthesiology, University Hospital of Basel
Locations (1):
- Department of Anaesthesiology, University Hospital of Basel (USB), Basel, Switzerland